CLINICAL TRIAL: NCT02149069
Title: Blood Management Program: Appropriateness of Transfusion Therapy in the Post - Operative Period.
Brief Title: Blood Management Program in the Post - Operative Period.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Principal Investigator, PAMELABERNI, Data Manager, Azienda USL Reggio Emilia - IRCCS
Other Study IDs: BMP - TRASFU1
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-06

CONDITIONS: Excessive Amount of Blood / Fluid Transfusion

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A care path in the field of transfusion medicine was creates at ASMN - IRCCS addressed to patients undergoing complex surgical procedures.

DETAILED DESCRIPTION:
This pathway is called Blood Management Program (BMP).

The implementation of this process should improve transfusion therapy in the peri-operative period in order to:

* correct the transfusional approach to surgical patients
* optimize the management of transfusional resources (red blood cells, plasma, platelets)
* optimize the management of plasma derivatives, drugs and techniques designed to limit the use of homologous blood

ELIGIBILITY:
Inclusion Criteria:

-All patients undergoing complex surgical procedures

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing complex surgical procedures
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of therapeutic appropriateness for Red Cells - Plasma - Platelets transfusion: comparison between prospective vs. retrospective data in ASMN ,Reggio Emilia (Italy) | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Erminia Di Bartolomeo, MD, Principal Investigator — ASMN-IRCCS
Locations (1):
- IRCCS-Arcispedale Santa Maria Nuova, Reggio Emilia, Emilia-Romagna, Italy